CLINICAL TRIAL: NCT04021628
Title: An Observational, Longitudinal, Natural History, Feasibility Cohort Study to Evaluate the Characteristics of Cytomegalovirus (CMV) Shedding in CMV Seropositive Women Throughout Pregnancy
Brief Title: Cytomegalovirus Shedding Characteristics in Pregnant Women
Acronym: cCHIPS
Status: Completed | Type: Observational
Sponsor: St George's, University of London (Other)
Collaborators: St George's University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2018.0296
Record Dates: First submitted 2019-07-01; First posted 2019-07-16 (Actual); Results first posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2023-12

CONDITIONS: CMV; Congenital Cmv; Maternal Infections Affecting Fetus or Newborn; Shedding Virus
Keywords: cmv; cytomegalovirus; shedding; excretion; congenital; cCMV; seropositive; maternal
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples with DNA of CMV virus, not human DNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention- not applicable — No intervention - not applicable

SUMMARY:
The cCHIPS study is a feasibility study for larger scale multi-centre studies and is designed as a single-centre observational cohort, longitudinal, natural history study.

The overarching aim of this study is to evaluate the feasibility of performing larger scale, multi-centre studies to evaluate the relationship between CMV shedding in pregnancy with congenital CMV (cCMV). There is no randomisation involved in this study and all participants will perform the same study procedures and receive treatment as usual.

The primary (main) objective is to evaluate the prevalence (percentage of occurrence) of CMV shedding in saliva, urine and vaginal secretions of CMV seropositive women throughout pregnancy.

The secondary objectives are to evaluate the quantity of CMV shedding in saliva, urine and vaginal secretions of CMV seropositive women throughout pregnancy, to compare the prevalence and quantity of CMV shedding in CMV seropositive women between different sources of shedding (saliva, urine or vaginal secretions) and different gestational stages, to identify risk factors for CMV shedding in CMV seropositive pregnant women, to evaluate the acceptability of the study procedures to the participating pregnant women, to evaluate the proportion of women approached who are recruited into the study and who are completing the study, and to evaluate the relationship between CMV specific cell mediated immunity (a type of immune protection following exposure to CMV) and CMV shedding in CMV seropositive pregnant women.

The tertiary objective is to compare the evaluation of CMV specific T cell immune responses (a type of CMV specific cell mediated immunity) between the two commercially available CMV-specific T cell immune response assays which are QuantiFERON-CMV and CMV-ELISPOT assays.

This study will aim to recruit 200 pregnant women.

This study will be undertaken in parallel with a separate study called RACE-FIT (REC reference number 18/SC/0360, IRAS ID 239977), which will have ethical approval to screen pregnant women with children less than 4 years of age booked for their antenatal care at St George's Hospital, London, identified during the antenatal combined screening bloods appointment or the antenatal booking appointment, for their CMV serology status on a sample of blood collected as part of the screening process. As part of the ethical approval sought for the RACE-FIT study and the cCHIPS study, the pregnant women screened and found to be CMV seronegative will be eligible for recruitment into the RACE-FIT study and those screened and found to be CMV seropositive will be eligible and approached for recruitment into the cCHIPS study.

The cCHIPS study aim to recruit over a 6 month period.

The study involves four visits (Visit 1, Visit 2, Visit 3, Visit 4) for each participant. The total study period for each participant will be between 6 to 8 months.

DETAILED DESCRIPTION:
The potential participants will be contacted via telephone, email and/or post by the study team. They will be screened for their eligibility, and if they are interested in participating, the first study visit (Visit 1) will be arranged where the written informed consent will be obtained then before any study related procedures.

Visit 1 will be held as soon as possible following screening, aiming up to 16 weeks and 6 days gestational age (early in pregnancy). Visit 2 will be aimed to coincide with the routine 20 gestational week appointment or any time in second trimester from 17 weeks and 0 days gestational age to 27 weeks and 6 days gestational age (middle of pregnancy). Visit 3 will be aimed to coincide with the routine 28 gestational week appointment or any time in the third trimester from 28 weeks and 0 days gestational age onwards (late in pregnancy), Visit 4 will be aimed to coincide with the participant's routine admission on the labour ward or postnatal ward after giving birth, or anytime from the time of birth to 1 week postnatal age (postpartum period).

At each study visit, the participants will be performing their own study samples of saliva, urine and vaginal secretions using the study specific self-sampling instructions provided. These self-samples will be tested for the presence and quantity of CMV DNA detected via a molecular technique called polymerase chain reaction (PCR). If consent is obtained, a blood sample will also be collected at each study visit to test for cellular mediated immunity. At the last visit, the participant will be offered to have her newborn baby tested for congenital CMV by collecting the newborn's saliva sample which will be tested for CMV DNA via PCR.

At each study visit, the participant will complete a short questionnaire on the participant's contact with their child(ren)'s saliva and urine (to identify risk factors for CMV shedding). At Visit 1, the participant will complete a background questionnaire (also to identify risk factors for CMV shedding)and at Visit 4 a feedback questionnaire (to assess feasibility).

Where possible the study visits and blood samples will be aimed to take place alongside the participants' routine antenatal appointments and routine blood tests respectively.

At the end of the study, up to 20 participants will be invited to take part in a process evaluation in the form of an interview by phone, skype or face to face to explore in depth the experiences of participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* CMV seropositive
* Willing and able to provide informed consent
* Living with child(ren), at least one of whom is less than four years old
* Willing to have saliva, urine and vaginal secretion sampling to be tested for CMV PCR
* Willing to be followed up until the postpartum period

Exclusion Criteria:

* Age less than 18 years
* Evidence of acute maternal CMV infection at the time of screening
* Documented immunodeficiency of any aetiology including the use of oral steroid therapy equivalent to >1mg/kg of prednisone per day for more than one week
* In the opinion of the investigator is unlikely to comply with the study procedures
* In the opinion of the investigator does not have adequate understanding or verbal and written English

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: CMV seropositive pregnant women with at least one child of less than four years of age
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shari Sapuan, Principal Investigator — St George's, University of London
Locations (1):
- St George's University Hospitals NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants Belonged to the Same Group: All participants belonged to the same group (non-interventional, observational cohort study)
Period: Overall Study
Arm/Group | All Participants Belonged to the Same Group
Started | 160 (Number of participants recruited at Visit 1)
Completed | 119 (Number of participants completed Visit 4 (last study visit))
Not Completed | 41

BASELINE CHARACTERISTICS:
Arm/Group | All Participants Belonged to the Same Group
Number analyzed (Participants) | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 160
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 160
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White British | 69
  Ethnicity: White Other | 39
  Ethnicity: South Asian | 23
  Ethnicity: Asian Other | 9
  Ethnicity: Black | 8
  Ethnicity: Mixed | 11
  Ethnicity: Other | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 160

OUTCOME MEASURES:

1. Primary Outcome: The Prevalence of CMV Shedding in Saliva, Urine and Vaginal Secretions of CMV Seropositive Women in Pregnancy
Description: The percentage of participants with detectable CMV virus (detected via polymerase chain reaction) in any bodily fluid (saliva, urine or vaginal secretions) at any point in pregnancy, and the percentage of participants with detectable CMV virus in each bodily fluid (saliva, urine and vaginal secretions) at any point in pregnancy.
Time Frame: 8 months
Population: The total number of participants with all complete data (no missing data)
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants Belonged to the Same Group
Number analyzed (Participants) | 123
Participants
  Prevalence in any bodily fluid | 27
  Prevalence in saliva | 4
  Prevalence in urine | 16
  Prevalence in vaginal secretions | 20

2. Secondary Outcome: The Proportion of CMV Shedding in Saliva, Urine and Vaginal Secretions of CMV Seropositive Women Throughout Pregnancy and Postpartum
Description: The proportion of detectable CMV virus (measured via polymerase chain reaction) in saliva, urine and vaginal secretions at individual study visits
Time Frame: 8 months
Measure: Count of Participants; unit: Participants
Groups:
- Visit 1 Saliva: Saliva sample (one per participant) tested for CMV DNA via PCR at Visit 1
- Visit 1 Urine: Urine sample (one per participant) tested for CMV DNA via PCR at Visit 1
- Visit 1 Vaginal Secretions: Vaginal secretions sample (one per participant) tested for CMV DNA via PCR at Visit 1
- Visit 2 Saliva: Saliva sample (one per participant) tested for CMV DNA via PCR at Visit 2
- Visit 2 Urine: Urine sample (one per participant) tested for CMV DNA via PCR at Visit 2
- Visit 2 Vaginal Secretions: Vaginal secretions sample (one per participant) tested for CMV DNA via PCR at Visit 2
- Visit 3 Saliva: Saliva sample (one per participant) tested for CMV DNA via PCR at Visit 3
- Visit 3 Urine: Urine sample (one per participant) tested for CMV DNA via PCR at Visit 3
- Visit 3 Vaginal Secretions: Vaginal secretions sample (one per participant) tested for CMV DNA via PCR at Visit 3
- Visit 4 Saliva: Saliva sample (one per participant) tested for CMV DNA via PCR at Visit 4
- Visit 4 Urine: Urine sample (one per participant) tested for CMV DNA via PCR at Visit 4
- Visit 4 Vaginal Secretions: Vaginal secretions sample (one per participant) tested for CMV DNA via PCR at Visit 4
Arm/Group | Visit 1 Saliva | Visit 1 Urine | Visit 1 Vaginal Secretions | Visit 2 Saliva | Visit 2 Urine | Visit 2 Vaginal Secretions | Visit 3 Saliva | Visit 3 Urine | Visit 3 Vaginal Secretions | Visit 4 Saliva | Visit 4 Urine | Visit 4 Vaginal Secretions
Number analyzed (Participants) | 155 | 155 | 156 | 141 | 141 | 142 | 134 | 136 | 135 | 102 | 111 | 83
Participants | 3 | 9 | 9 | 3 | 10 | 10 | 3 | 9 | 10 | 0 | 7 | 5

3. Secondary Outcome: The Quantity of CMV Shedding in Saliva, Urine and Vaginal Secretions in CMV Seropositive Women Throughout Pregnancy and Postpartum
Description: The quantity of detectable CMV virus (measured via quantitative polymerase chain reaction in IU/ml) in saliva, urine and vaginal secretions at individual study visits
Time Frame: 8 months
Population: As there was no CMV DNA via PCR detected from the participants' saliva samples tested at Visit 4, this arm was excluded from the statistical analysis. Where CMV DNA was detected below the assay's limit of quantification, the quantity was defined as 1.0 IU/ml for the purpose of statistical analysis.
Measure: Median (Full Range); unit: IU/ml
Groups:
- Visit 1 Saliva: Saliva sample (one per participant) tested for CMV DNA via PCR at Visit 1 (up to 16 weeks and 6 days gestational age)
- Visit 1 Urine: Urine sample (one per participant) tested for CMV DNA via PCR at Visit 1 (up to 16 weeks and 6 days gestational age)
- Visit 1 Vaginal Secretions: Vaginal secretions sample (one per participant) tested for CMV DNA via PCR at Visit 1 (up to 16 weeks and 6 days gestational age)
- Visit 2 Saliva: Saliva sample (one per participant) tested for CMV DNA via PCR at Visit 2 (from 17 weeks and 0 days gestational age to 27 weeks and 6 days gestational age)
- Visit 2 Urine: Urine sample (one per participant) tested for CMV DNA via PCR at Visit 2 (from 17 weeks and 0 days gestational age to 27 weeks and 6 days gestational age)
- Visit 2 Vaginal Secretions: Vaginal secretions sample (one per participant) tested for CMV DNA via PCR at Visit 2 (from 17 weeks and 0 days gestational age to 27 weeks and 6 days gestational age)
- Visit 3 Saliva: Saliva sample (one per participant) tested for CMV DNA via PCR at Visit 3 (from 28 weeks and 0 days gestational age onwards)
- Visit 3 Urine: Urine sample (one per participant) tested for CMV DNA via PCR at Visit 3 (from 28 weeks and 0 days gestational age onwards)
- Visit 3 Vaginal Secretions: Vaginal secretions sample (one per participant) tested for CMV DNA via PCR at Visit 3 (from 28 weeks and 0 days gestational age onwards)
- Visit 4 Urine: Urine sample (one per participant) tested for CMV DNA via PCR at Visit 4 (anytime from the time of birth to 1 week postnatal age)
- Visit 4 Vaginal Secretions: Vaginal secretions sample (one per participant) tested for CMV DNA via PCR at Visit 4 (anytime from the time of birth to 1 week postnatal age)
Arm/Group | Visit 1 Saliva | Visit 1 Urine | Visit 1 Vaginal Secretions | Visit 2 Saliva | Visit 2 Urine | Visit 2 Vaginal Secretions | Visit 3 Saliva | Visit 3 Urine | Visit 3 Vaginal Secretions | Visit 4 Urine | Visit 4 Vaginal Secretions
Number analyzed (Participants) | 3 | 9 | 9 | 3 | 10 | 10 | 3 | 9 | 10 | 7 | 5
IU/ml | 521.0 [227.0 to 689.0] | 1.0 [1.0 to 10900.0] | 800.0 [132.0 to 32000.0] | 693.0 [402.0 to 768.0] | 104.5 [1.0 to 4930.0] | 189.5 [1.0 to 7500.0] | 539.0 [137.0 to 634.0] | 1.0 [1.0 to 373.0] | 640.5 [106.0 to 6480.0] | 1.0 [1.0 to 2490.0] | 260.0 [166.0 to 639.0]

4. Secondary Outcome: The Proportion of Pregnant Women Approached Who Are Recruited Into the Study
Description: The percentage of women approached who are then recruited into the study
Time Frame: 8 months
Measure: Count of Participants; unit: Participants
Groups:
- Proportion of Women Approached Who Were Eligible for Screening: Pregnant women who were approached at early antenatal appointment and were found to be eligible for screening
- Proportion of Eligible Approached Women Who Had Screening: Pregnant women who were approached and found to be eligible for screening
- Proportion of Screened Women Eligible for Recruitment: Pregnant women who were screened and found to be eligible for recruitment
- Proportion of Eligible Screened Women Who Were Recruited: Pregnant women who were recruited from those screened and eligible for recruitment
Arm/Group | Proportion of Women Approached Who Were Eligible for Screening | Proportion of Eligible Approached Women Who Had Screening | Proportion of Screened Women Eligible for Recruitment | Proportion of Eligible Screened Women Who Were Recruited
Number analyzed (Participants) | 3339 | 966 | 804 | 384
Participants | 966 | 804 | 384 | 160

5. Secondary Outcome: The Proportion of Participating Pregnant Women Completing the Study
Time Frame: 8 months
Measure: Count of Participants; unit: Participants
Groups:
- The Proportion of Participants Who Completed All Study Visits: The percentage of participants who completed all study visits (provide urine, saliva and vaginal secretion samples at all four study visits)
- The Proportion of Participants Who Completed All Study Visits During Pregnancy: The percentage of participants who completed Visit 1, Visit 2 and Visit 3 (provide urine, saliva and vaginal secretion samples at Visit 1, Visit 2 and Visit 3)
- The Proportion of Participants Who Completed the Last Study Visit: The percentage of participants who completed Visit 1 and Visit 4, regardless of whether Visit 2 or Visit 3 were completed
Arm/Group | The Proportion of Participants Who Completed All Study Visits | The Proportion of Participants Who Completed All Study Visits During Pregnancy | The Proportion of Participants Who Completed the Last Study Visit
Number analyzed (Participants) | 160 | 160 | 160
Participants | 66 | 123 | 119

6. Secondary Outcome: The Acceptability of the Study Procedures to Participating Pregnant Women
Description: Descriptive summary of the mean scores of each feedback statement (scale 1 to 5, where higher score was indicative of higher agreement to the feedback statement) from the Feedback Questionnaire completed by participants at the last study visit
Time Frame: 8 months
Population: Total number of participant who completed the Feedback Questionnaire at Visit 4 (last study visit)
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Groups:
- Language and Information of the Study Poster Was Just Right; Happy to be Approached by Study Team at Routine Antenatal Appointment; Language and Information on the Screening Invitation Letter Was Just Right; Happy to Ask Study Team Questions at Screening Which Were Appropriately Addressed; Satisfied With Information Received at Screening and Understood Next Steps; Language and Information on Screening Results and Study Invitation Letter Was Just Right; Happy to Contact Study Team After Receiving the Letter on Screening Results and Study Invitation; Happy for Study Team to Contact After Receiving the Letter on Screening Results and Study Invitation; Happy to Ask Questions (and Addressed), and With Information About Recruitment Visit on the Phone; Language and Information in Participant Information Sheet Was Just Right; Happy to Complete All Procedures at Recruitment Visit (Visit 1); Happy to Ask Questions at Recruitment Visit (Visit 1) Which Were Appropriately Addressed; Satisfied With Information Received at Recruitment Visit (Visit 1) and Understood Next Steps; Willing to Complete the Background Questionnaire; Willing to Complete the Contact Questionnaire at All Study Visits; The Self-sampling Written Instructions Were Simple and Clear; Willing to Perform Self-sampling of Saliva Samples for All Study Visits; Willing to Perform Self-sampling of Urine Samples for All Study Visits; Willing to Perform Self-sampling of Vaginal Secretions for All Study Visits; Willing to Perform All Self-sampling for All Study Visits; Willing to Have Blood Samples Taken for All Study Visits; Willing to Have Additional Blood Samples Taken on Top of Routine Antenatal Blood Samples; Happy to Have the Option to Test Newborn for Congenital CMV; Willing to be Part of All Four Study Visits; Study Visit Timeline Was Not Troublesome; Happy to Receive Study Visit Text Reminders; Willing to Attend Study Visits That do Not Coincide With Routine Antenatal Appoinments; Prefer to Have Study Visits at the Same Time as Routine Antenatal Appointments; Prefer to Have Study Visits at Home; Willing to Contact Study Team When in Labour or Soon After Birth; Willing to Have Study Visit Soon After Birth Whilst Still in Hospital; Willing to Have Study Visit With Newborn in Hospital/Clinic After Already Being Discharged Home: Feedback statement from the Feedback Questionnaire. Score between 1 to 5, where higher score indicated higher agreement to the feedback statement.
Arm/Group | Language and Information of the Study Poster Was Just Right | Happy to be Approached by Study Team at Routine Antenatal Appointment | Language and Information on the Screening Invitation Letter Was Just Right | Happy to Ask Study Team Questions at Screening Which Were Appropriately Addressed | Satisfied With Information Received at Screening and Understood Next Steps | Language and Information on Screening Results and Study Invitation Letter Was Just Right | Happy to Contact Study Team After Receiving the Letter on Screening Results and Study Invitation | Happy for Study Team to Contact After Receiving the Letter on Screening Results and Study Invitation | Happy to Ask Questions (and Addressed), and With Information About Recruitment Visit on the Phone | Language and Information in Participant Information Sheet Was Just Right | Happy to Complete All Procedures at Recruitment Visit (Visit 1) | Happy to Ask Questions at Recruitment Visit (Visit 1) Which Were Appropriately Addressed | Satisfied With Information Received at Recruitment Visit (Visit 1) and Understood Next Steps | Willing to Complete the Background Questionnaire | Willing to Complete the Contact Questionnaire at All Study Visits | The Self-sampling Written Instructions Were Simple and Clear | Willing to Perform Self-sampling of Saliva Samples for All Study Visits | Willing to Perform Self-sampling of Urine Samples for All Study Visits | Willing to Perform Self-sampling of Vaginal Secretions for All Study Visits | Willing to Perform All Self-sampling for All Study Visits | Willing to Have Blood Samples Taken for All Study Visits | Willing to Have Additional Blood Samples Taken on Top of Routine Antenatal Blood Samples | Happy to Have the Option to Test Newborn for Congenital CMV | Willing to be Part of All Four Study Visits | Study Visit Timeline Was Not Troublesome | Happy to Receive Study Visit Text Reminders | Willing to Attend Study Visits That do Not Coincide With Routine Antenatal Appoinments | Prefer to Have Study Visits at the Same Time as Routine Antenatal Appointments | Prefer to Have Study Visits at Home | Willing to Contact Study Team When in Labour or Soon After Birth | Willing to Have Study Visit Soon After Birth Whilst Still in Hospital | Willing to Have Study Visit With Newborn in Hospital/Clinic After Already Being Discharged Home
Number analyzed (Participants) | 58 | 58 | 58 | 58 | 58 | 58 | 58 | 58 | 58 | 58 | 58 | 58 | 58 | 58 | 58 | 58 | 58 | 58 | 58 | 58 | 58 | 58 | 58 | 58 | 58 | 58 | 58 | 58 | 58 | 58 | 58 | 58
Score on a scale | 4.03 [3.80 to 4.27] | 4.57 [4.32 to 4.82] | 4.38 [4.11 to 4.65] | 4.48 [4.23 to 4.74] | 4.50 [4.29 to 4.76] | 4.22 [3.98 to 4.47] | 3.98 [3.72 to 4.24] | 4.43 [4.18 to 4.68] | 4.52 [4.26 to 4.77] | 4.45 [4.22 to 4.68] | 4.55 [4.30 to 4.80] | 4.59 [4.33 to 4.84] | 4.57 [4.34 to 4.80] | 4.64 [4.39 to 4.88] | 4.62 [4.38 to 4.87] | 4.53 [4.31 to 4.76] | 4.71 [4.47 to 4.95] | 4.64 [4.39 to 4.89] | 4.26 [3.94 to 4.58] | 4.40 [4.13 to 4.67] | 4.36 [4.10 to 4.62] | 4.16 [3.87 to 4.44] | 4.52 [4.27 to 4.76] | 4.71 [4.48 to 4.93] | 4.59 [4.37 to 4.80] | 4.74 [4.52 to 4.96] | 3.31 [2.99 to 3.63] | 4.62 [4.36 to 4.88] | 3.22 [2.98 to 3.47] | 4.09 [3.82 to 4.36] | 4.38 [4.15 to 4.60] | 3.14 [2.85 to 3.42]

7. Secondary Outcome: The Association of Demographics With CMV Shedding in CMV Seropositive Women in Pregnancy
Description: The multiple logistic regression of CMV shedding as an outcome (dependent variable; detected or not detected) at any visit during pregnancy with demographic factors (independent variable) as a predictor, adjusted for all demographic variables described, using odds ratio in the results between CMV seropositive women with CMV shedding and without CMV shedding, with 95% confidence interval.
Time Frame: 8 months
Population: Multiple logistic regression with CMV shedding in pregnancy status (detected or not detected) as the dependent variable (outcome) and the demographic variables as the independent variables (predictors), on participants where all saliva, urine and vaginal secretion samples were collected and tested at Visit 1, Visit 2 and Visit 3.
Measure: Number (95% Confidence Interval); unit: Odds Ratio
Groups:
- CMV Shedding Detected at Any Point in Pregnancy in CMV-seropositive Women: Participants with at least one occasion of CMV shedding detected in saliva, urine or vaginal secretion samples at Visit 1(up to 16 weeks and 6 days gestational age), Visit 2 (from 17 weeks and 0 days gestational age to 27 weeks and 6 days gestational age) or Visit 3 (from 28 weeks and 0 days gestational age onwards). All three sample types must have been collected and tested at all three visit types.
Arm/Group | CMV Shedding Detected at Any Point in Pregnancy in CMV-seropositive Women
Number analyzed (Participants) | 123
Odds Ratio
  Age group (<30y,30-39y,>39) | 3.17 [0.89 to 11.34]
  Ethnicity (White(W)British,WOther(O),SouthAsian(A),AO,Black,Mixed,O) | 0.95 [0.62 to 1.47]
  Born in UK (Yes, No) | 1.02 [0.67 to 3.93]
  Duration in UK (<5yrs,5-15yrs,>15yrs) | 1.41 [0.52 to 3.80]
  Highest Education (PhD/Masters, Degree, Diploma, ALevels/GCSE) | 0.99 [0.60 to 1.63]
  Total pregnancies (2,3,>3) | 0.36 [0.16 to 0.81]
  No. of children (1,2,>2): OR 2.0 [95% CI 0.3,12.3], p=0.445 | 2.73 [0.63 to 11.82]
  Work regularly with children (yes,no) | 1.60 [0.47 to 5.46]
  No. of households (<=3,>3) | 0.91 [0.20 to 4.16]
  No. of people per bedroom (1,2,3) | 0.73 [0.21 to 2.56]

8. Secondary Outcome: The Association of Contact With Young Children's Bodily Fluids With CMV Shedding in CMV Seropositive Women Throughout Pregnancy and Postpartum
Description: The association between CMV shedding detection and the specific types of contact with child(ren)'s bodily fluids as assessed in the contact questionnaire at each visit, performed using logistic regression (CMV shedding detection as the outcome variable, the specific types of contact with children's bodily fluids as the predictor varible), adjusted for age, ethnicity, education, and amount of children, with the detection of shedding as a binary outcome, using odds ratio in the results between CMV-seropositive with CMV shedding and without CMV shedding, with 95% confidence intervals.
Time Frame: 8 months
Population: The association between CMV shedding detection and the specific types of contact with child(ren)'s bodily fluids as assessed in the contact questionnaire at each visit, performed using adjusted logistic regression.
Measure: Number (95% Confidence Interval); unit: Adjusted Odds Ratio
Groups:
- Visit 1 (up to 16 Weeks and 6 Days Gestational Age); Visit 2 (From 17 Weeks and 0 Days Gestational Age to 27 Weeks and 6 Days Gestational Age): Likert scale survey (out to 5) on specific types of hygiene-based contact with child(ren)'s bodily fluids
- Visit 3 (From 28 Weeks and 0 Days Gestational Age Onwards): Likert scale survey (out to 5) on specific types of hygiene-based contact with child(ren)'s bodily fluids (from 28 weeks and 0 days gestational age onwards)
- Visit 4 (Anytime From the Time of Birth to 1 Week Postnatal Age): Likert scale survey (out to 5) on specific types of hygiene-based contact with child(ren)'s bodily fluids (anytime from the time of birth to 1 week postnatal age)
Arm/Group | Visit 1 (up to 16 Weeks and 6 Days Gestational Age) | Visit 2 (From 17 Weeks and 0 Days Gestational Age to 27 Weeks and 6 Days Gestational Age) | Visit 3 (From 28 Weeks and 0 Days Gestational Age Onwards) | Visit 4 (Anytime From the Time of Birth to 1 Week Postnatal Age)
Number analyzed (Participants) | 152 | 119 | 111 | 52
Adjusted Odds Ratio
  Wash hands with soap after handling child's faeces | 0 [0 to 0] | 0.74 [0.40 to 1.40] | 0.74 [0.35 to 1.57] | 0.99 [0.27 to 3.69]
  Wash hands without soap after handling child's faeces | 0.81 [0.45 to 1.46] | 1.10 [0.70 to 1.74] | 1.22 [0.76 to 1.95] | 1.04 [0.44 to 2.46]
  Clean hands with alcohol gel after handling child's faeces | 1.23 [0.70 to 2.16] | 0.94 [0.55 to 1.62] | 1.49 [0.88 to 2.51] | 0.54 [0.20 to 1.45]
  Wash hands with soap after handling with child's urine | 1.23 [0.62 to 2.43] | 0.90 [0.51 to 1.56] | 0.47 [0.26 to 0.85] | 0.99 [0.35 to 2.79]
  Wash hands without soap after handling with child's urine | 0.72 [0.41 to 1.28] | 0.84 [0.51 to 1.38] | 1.16 [0.68 to 1.98] | 1.29 [0.57 to 2.92]
  Clean hands with alcohol gel after handling with child's urine | 1.25 [0.74 to 2.09] | 1.21 [0.70 to 2.09] | 1.34 [0.76 to 2.35] | 0.69 [0.25 to 1.91]
  Wash hands with soap after wiping child's nose | 1.47 [0.80 to 2.71] | 1.58 [0.90 to 2.78] | 0.54 [0.26 to 1.12] | 2.19 [0.72 to 6.68]
  Wash hands without soap after wiping child's nose | 1.08 [0.60 to 1.92] | 0.73 [0.40 to 1.35] | 0.62 [0.27 to 1.34] | 1.57 [0.68 to 3.63]
  Clean hands with alcohol gel after wiping child's nose | 1.50 [0.78 to 2.89] | 0.93 [0.49 to 1.77] | 0.84 [0.40 to 1.79] | 0.31 [0.07 to 1.43]
  Put child's dummy in own mouth | 1.09 [0.69 to 1.74] | 1.00 [0.59 to 1.70] | 1.17 [0.66 to 2.09] | 0 [0 to 0]
  Eat child's leftover food | 0.57 [0.33 to 0.98] | 1.16 [0.69 to 1.98] | 0.77 [0.42 to 1.42] | 2.14 [0.67 to 6.78]
  Eat with child's used cutlery | 0.64 [0.36 to 1.12] | 1.14 [0.71 to 1.84] | 1.01 [0.60 to 1.72] | 0.67 [0.25 to 1.81]
  Drink from child's used cup | 0.55 [0.31 to 0.99] | 0.78 [0.46 to 1.31] | 0.84 [0.50 to 1.43] | 0.70 [0.28 to 1.77]
  Kiss child on the lips | 0.87 [0.55 to 1.37] | 1.22 [0.77 to 1.93] | 1.23 [0.73 to 2.08] | 1.06 [0.53 to 2.10]

9. Secondary Outcome: The Prevalence of CMV-specific T-cell Immune Responses as Measured by CMV-QuantiFERON in CMV Seropositive Women in Pregnancy
Description: The percentage of the number of participants with positive CMV-QuantiFERON results over the total number of participants tested with CMV-QuantiFERON at any point in pregnancy
Time Frame: 8 months
Population: Not all participant recruited in the study were tested with CMV -QuantiFERON assay.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants Belonged to the Same Group
Number analyzed (Participants) | 88
Participants | 62

10. Secondary Outcome: The Prevalence of CMV-specific T-cell Immune Responses as Measured by CMV-ELISPOT in CMV Seropositive Women in Pregnancy
Description: The percentage of the number of participants with responsive CMV-ELISPOT results over the total number of participants tested with CMV-ELISPOT at any point in pregnancy
Time Frame: 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants Belonged to the Same Group
Number analyzed (Participants) | 67
Participants | 67

11. Secondary Outcome: The Proportion of CMV-specific T-cell Immune Responses as Measured by CMV-QuantiFERON in CMV Seropositive Women Throughout Pregnancy and Postpartum
Description: The percentage of the number of participants with positive CMV-QuantiFERON results over the total number of participants tested for CMV-QuantiFERON at each study visit
Time Frame: 8 months
Measure: Count of Participants; unit: Participants
Groups:
- Proportion of Participants With Positive CMV QuantiFERON Results at Visit 1: Participants with positive CMV QuantiFERON results at Visit 1 over the total number of participants tested for CMV-QuantiFERON at Visit 1 (up to 16 weeks and 6 days gestational age)
- Proportion of Participants With Positive CMV QuantiFERON Results at Visit 2: Participants with positive CMV QuantiFERON results at Visit 2 over the total number of participants tested for CMV-QuantiFERON at Visit 2 (from 17 weeks and 0 days gestational age to 27 weeks and 6 days gestational age)
- Proportion of Participants With Positive CMV QuantiFERON Results at Visit 3: Participants with positive CMV QuantiFERON results at Visit 3 over the total number of participants tested for CMV-QuantiFERON at Visit 3 (from 28 weeks and 0 days gestational age onwards)
- Proportion of Participants With Positive CMV QuantiFERON Results at Visit 4: Participants with positive CMV QuantiFERON results at Visit 4 over the total number of participants tested for CMV-QuantiFERON at Visit 4 (anytime from the time of birth to 1 week postnatal age)
Arm/Group | Proportion of Participants With Positive CMV QuantiFERON Results at Visit 1 | Proportion of Participants With Positive CMV QuantiFERON Results at Visit 2 | Proportion of Participants With Positive CMV QuantiFERON Results at Visit 3 | Proportion of Participants With Positive CMV QuantiFERON Results at Visit 4
Number analyzed (Participants) | 72 | 52 | 42 | 16
Participants | 50 | 39 | 31 | 10

12. Secondary Outcome: The Proportion of CMV-specific T-cell Immune Responses as Measured by CMV-ELISPOT in CMV Seropositive Women Throughout Pregnancy and Postpartum
Description: The percentage of the number of participants with responsive CMV-ELISPOT results (a positive spot count to IE-1 and/or pp65 antigen) over the total number of participants tested for CMV-ELISPOT at each study visit
Time Frame: 8 months
Measure: Count of Participants; unit: Participants
Groups:
- The Proportion of Participants With Responsive CMV-ELISPOT at Visit 1: The percentage of participants with responsive CMV-ELISPOT results (a positive spot count to IE-1 and/or pp65 antigen) at Visit 1 over the number of participants with CMV-ELISPOT tested at Visit 1(up to 16 weeks and 6 days gestational age)
- The Proportion of Participants With Responsive CMV-ELISPOT Results at Visit 2: The percentage of participants with responsive CMV-ELISPOT results (a positive spot count to IE-1 and/or pp65 antigen) at Visit 2 over the number of participants with CMV-ELISPOT tested at Visit 2 (from 17 weeks and 0 days gestational age to 27 weeks and 6 days gestational age)
- The Proportion of Participants With Responsive CMV-ELISPOT Results at Visit 3: The percentage of participants with responsive CMV-ELISPOT results (a positive spot count to IE-1 and/or pp65 antigen) at Visit 3 over the number of participants with CMV-ELISPOT tested at Visit 3 (from 28 weeks and 0 days gestational age onwards)
- The Proportion of Participants With Responsive CMV-ELISPOT Results at Visit 4: The percentage of participants with responsive CMV-ELISPOT results (a positive spot count to IE-1 and/or pp65 antigen) at Visit 4 over the number of participants with CMV-ELISPOT tested at Visit 4 (anytime from the time of birth to 1 week postnatal age)
Arm/Group | The Proportion of Participants With Responsive CMV-ELISPOT at Visit 1 | The Proportion of Participants With Responsive CMV-ELISPOT Results at Visit 2 | The Proportion of Participants With Responsive CMV-ELISPOT Results at Visit 3 | The Proportion of Participants With Responsive CMV-ELISPOT Results at Visit 4
Number analyzed (Participants) | 49 | 25 | 26 | 8
Participants | 49 | 24 | 25 | 8

13. Secondary Outcome: The Association Between CMV-specific T Cell Immune Response and CMV Shedding in CMV Seropositive Pregnant Women as Measured by CMV-QuantiFERON
Description: The logistic regression of CMV shedding as an outcome (dependent variable; detected or not detected) at a visit with CMV-QuantiFERON assay results (independent variable; positive or negative) as a predictor at the reciprocal visit, adjusted for age and ethnicity, using odds ratio in the results between CMV seropositive women with CMV shedding and without CMV shedding, with 95% confidence interval.
Time Frame: 8 months
Population: The logistic regression of CMV shedding as an outcome (dependent variable; detected or not detected) at a visit with CMV-QuantiFERON assay results (independent variable; positive or negative) as a predictor at the reciprocal visit, adjusted for age and ethnicity, in CMV seropositive women.
Measure: Number (95% Confidence Interval); unit: Odds Ratio
Groups:
- Visit 1: Outcome of CMV Shedding Using CMV QuantiFERON Results as Predictor: The logistic regression of CMV shedding as an outcome (dependent variable; detected or not detected) at Visit 1 (up to 16 weeks and 6 days gestational age )with CMV QuantiFERON assay results (independent variable; positive or negative) as a predictor at the reciprocal visit, adjusted for age and ethnicity, in CMV seropositive women.
- Visit 2: Outcome of CMV Shedding Using CMV QuantiFERON Results as Predictor: The logistic regression of CMV shedding as an outcome (dependent variable; detected or not detected) at Visit 2 (from 17 weeks and 0 days gestational age to 27 weeks and 6 days gestational age) with CMV QuantiFERON assay results (independent variable; positive or negative) as a predictor at the reciprocal visit, adjusted for age and ethnicity, in CMV seropositive women.
- Visit 3: Outcome of CMV Shedding Using CMV QuantiFERON Results as Predictor: The logistic regression of CMV shedding as an outcome (dependent variable; detected or not detected) at Visit 3 (from 28 weeks and 0 days gestational age onwards) with CMV QuantiFERON assay results (independent variable; positive or negative) as a predictor at the reciprocal visit, adjusted for age and ethnicity, in CMV seropositive women.
- Visit 4: Outcome of CMV Shedding Using CMV QuantiFERON Results as Predictor: The logistic regression of CMV shedding as an outcome (dependent variable; detected or not detected) at Visit 4 (anytime from the time of birth to 1 week postnatal age) with CMV QuantiFERON assay results (independent variable; positive or negative) as a predictor at the reciprocal visit, adjusted for age and ethnicity, in CMV seropositive women.
Arm/Group | Visit 1: Outcome of CMV Shedding Using CMV QuantiFERON Results as Predictor | Visit 2: Outcome of CMV Shedding Using CMV QuantiFERON Results as Predictor | Visit 3: Outcome of CMV Shedding Using CMV QuantiFERON Results as Predictor | Visit 4: Outcome of CMV Shedding Using CMV QuantiFERON Results as Predictor
Number analyzed (Participants) | 72 | 51 | 42 | 12
Odds Ratio | 0.56 [0.11 to 2.76] | 1.19 [0.21 to 6.68] | 2.82 [0.26 to 30.66] | 0.00 [0.00 to 0.00]

14. Secondary Outcome: The Association Between CMV-specific T Cell Immune Response and CMV Shedding in CMV Seropositive Pregnant Women as Measured by CMV-ELISPOT
Description: The logistic regression of CMV shedding as an outcome (dependent variable; detected or not detected) at a visit with CMV-ELISPOT assay results (independent variable; spot count) as a predictor at the reciprocal visit, adjusted for age and ethnicity, using odds ratio in the results between CMV seropositive women with CMV shedding and without CMV shedding, with 95% confidence interval.
Time Frame: 8 months
Population: The logistic regression of CMV shedding as an outcome (dependent variable; detected or not detected) at a visit with CMV-ELISPOT assay results (independent variable; spot count) as a predictor at the reciprocal visit, adjusted for age and ethnicity, in CMV seropositive women.
Measure: Number (95% Confidence Interval); unit: Odds Ratio
Groups:
- Visit 1: Outcome of CMV Shedding With CMV ELISPOT IE-1 Spot Count as the Predictor: The logistic regression of CMV shedding as an outcome (dependent variable; detected or not detected) at Visit 1 (up to 16 weeks and 6 days gestational age) with CMV-ELISPOT IE-1 assay results (independent variable; spot count) as a predictor at the reciprocal visit, adjusted for age and ethnicity, in CMV seropositive women.
- Visit 1: Outcome of CMV Shedding With CMV ELISPOT pp65 Spot Count as the Predictor: The logistic regression of CMV shedding as an outcome (dependent variable; detected or not detected) at Visit 1 (up to 16 weeks and 6 days gestational age) with CMV-ELISPOT pp65 assay results (independent variable; spot count) as a predictor at the reciprocal visit, adjusted for age and ethnicity, in CMV seropositive women.
- Visit 2: Outcome of CMV Shedding With CMV-ELISPOT IE-1 Spot Count as the Predictor: The logistic regression of CMV shedding as an outcome (dependent variable; detected or not detected) at Visit 2 (from 17 weeks and 0 days gestational age to 27 weeks and 6 days gestational age) with CMV-ELISPOT IE-1 assay results (independent variable; spot count) as a predictor at the reciprocal visit, adjusted for age and ethnicity, in CMV seropositive women.
- Visit 2: Outcome of CMV Shedding With CMV-ELISPOT pp65 Spot Count as the Predictor: The logistic regression of CMV shedding as an outcome (dependent variable; detected or not detected) at Visit 2 (from 17 weeks and 0 days gestational age to 27 weeks and 6 days gestational age) with CMV-ELISPOT pp65 assay results (independent variable; spot count) as a predictor at the reciprocal visit, adjusted for age and ethnicity, in CMV seropositive women.
- Visit 3: Outcome of CMV Shedding With CMV-ELISPOT IE-1 Spot Count as the Predictor: The logistic regression of CMV shedding as an outcome (dependent variable; detected or not detected) at Visit 3 (from 28 weeks and 0 days gestational age onwards) with CMV-ELISPOT IE-1 assay results (independent variable; spot count) as a predictor at the reciprocal visit, adjusted for age and ethnicity, in CMV seropositive women.
- Visit 3: Outcome of CMV Shedding With CMV-ELISPOT pp65 Spot Count as the Predictor: The logistic regression of CMV shedding as an outcome (dependent variable; detected or not detected) at Visit 3 (from 28 weeks and 0 days gestational age onwards) with CMV-ELISPOT pp65 assay results (independent variable; spot count) as a predictor at the reciprocal visit, adjusted for age and ethnicity, in CMV seropositive women.
Arm/Group | Visit 1: Outcome of CMV Shedding With CMV ELISPOT IE-1 Spot Count as the Predictor | Visit 1: Outcome of CMV Shedding With CMV ELISPOT pp65 Spot Count as the Predictor | Visit 2: Outcome of CMV Shedding With CMV-ELISPOT IE-1 Spot Count as the Predictor | Visit 2: Outcome of CMV Shedding With CMV-ELISPOT pp65 Spot Count as the Predictor | Visit 3: Outcome of CMV Shedding With CMV-ELISPOT IE-1 Spot Count as the Predictor | Visit 3: Outcome of CMV Shedding With CMV-ELISPOT pp65 Spot Count as the Predictor
Number analyzed (Participants) | 49 | 49 | 24 | 24 | 26 | 26
Odds Ratio | 1.00 [0.99 to 1.01] | 0.99 [0.98 to 1.00] | 1.00 [0.99 to 1.00] | 0.97 [0.94 to 0.99] | 1.00 [0.98 to 1.01] | 0.99 [0.98 to 1.01]

ADVERSE EVENTS:
Time Frame: 8 months
Description: The definitions and assessment of adverse event and serious adverse event are in accordance with the Health Research Authority, England, United Kingdom
Arm/Group | All Participants Belonged to the Same Group
All-Cause Mortality (participants affected / at risk) | 0/160
Serious Adverse Events (participants affected / at risk) | 11/160
Other Adverse Events (participants affected / at risk) | 11/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants Belonged to the Same Group (N=160)
Postpartum haemorrhage requiring blood transfusion (Reproductive system and breast disorders) | 4 (4)
Admission of newborn to neonatal unit (Reproductive system and breast disorders) | 7 (7)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants Belonged to the Same Group (N=160)
Emergency caesarian section (Reproductive system and breast disorders) | 1 (1)
Gestational diabetes (Reproductive system and breast disorders) | 7 (7)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Induction of labour for IUGR (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-25): https://cdn.clinicaltrials.gov/large-docs/28/NCT04021628/Prot_SAP_000.pdf